CLINICAL TRIAL: NCT00033137
Title: Birt-Hogg-Dub(SqrRoot)(Copyright) Syndrome: Characterization of the FLCN Disease Gene and Predisposition to Renal Cancer, Cutaneous Fibrofolliculoma and Pulmonary Cysts
Brief Title: Genetic Analysis of Birt Hogg-Dube Syndrome and Characterization of Predisposition to Kidney Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020159; 02-C-0159; NCT00039533 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Kidney Neoplasms; Kidney Cancer; Pneumothorax; FLCN Protein, Human
Keywords: Pneumothorax; Kidney; Fibrofolliculoma; BHD; Neoplasms; Natural History
MeSH Terms: conditions — Kidney Neoplasms; Pneumothorax; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Family Members: A relative of a patient with a confirmed or suspected diagnosis of BHD (related by blood)
- Non-Biologic Family Members: Spouses enrolled primarily for linkage analysis(Spouses have been removed from the inclusion criteria for this study. This closed cohort has been created for spouses previously enrolled on study.)
- Patients: Patients with phenotype or genotype suggestive of Birt Hogg Dub(SqrRoot)(Copyright) and/or Renal tumor histology consistent with BHD

SUMMARY:
This study will investigate the genetic cause of Birt Hogg-Dube (BHD) syndrome and the relationship of this disorder to kidney cancer. BHD is a rare inherited condition characterized by papules, or bumps-benign tumors involving hair follicles-on the head and neck. People with BHD are at increased risk of developing kidney cancer. Scientists have identified the chromosome (strand of genetic material in the cell nucleus) that contains the BHD gene and the region of the gene on the chromosome. This study will try to learn more about:

* The characteristics and type of kidney tumors associated with BHD
* The risk of kidney cancer in people with BHD
* Whether more than one gene causes BHD
* The genetic mutations (changes) responsible for BHD

Patients with known or suspected Birt Hogg-Dube syndrome, and their family members, may be eligible for this study. Candidates will be screened with a family history and review of medical records, including pathology reports for tumors, and films of computed tomography (CT) and magnetic resonance imaging (MRI) scans.

Participants may undergo various tests and procedures, including the following:

* Physical examination
* Review of personal and family history with a cancer doctor, cancer nurses, kidney surgeon, and genetic counselor
* Chest and other x-rays
* Ultrasound (imaging study using sound waves)
* MRI (imaging study using radiowaves and a magnetic field)
* CT scans of the chest and abdomen (imaging studies using radiation)
* Blood tests for blood chemistries and genetic testing
* Skin evaluation, including a skin biopsy (surgical removal of a small skin tissue sample for microscopic evaluation)
* Cheek swab or mouthwash to collect cells for genetic analysis
* Lung function studies
* Medical photography of skin lesions

These tests will be done on an outpatient basis in either one day or over 3 to 4 days. When the studies are complete, participants will receive counseling about the findings and recommendations. Patients with kidney lesions may be asked to return periodically, such as every 3 to 36 months, based on their individual condition, to document the rate of progression of the lesions.

DETAILED DESCRIPTION:
Background:

* Birt-Hogg-Dube (BHD) is a rare, autosomal dominantly inherited disorder which confers susceptibility to develop multifocal, bilateral renal cancer, spontaneous pneumothorax and fibrofolliculomas.
* BHD is caused by mutations in the FLCN gene located on Chromosome17p11.2
* Defining the genetic and biochemical pathways leading to renal tumorigenesis in BHD may lead to the development of new molecularly targeted drugs.

Objectives:

* To define the types and characteristics (including patterns of growth) of renal cancer associated with BHD
* To determine the risk of renal cancer, lung cysts and fibrofolliculomas in individuals with BHD
* To define the natural history of BHD related renal tumors
* To determine if other genes contribute to BHD
* Identify genotype/phenotype correlations

Eligibility:

* Individuals suspected or known to have phenotype or genotype suggestive of Birt-Hogg-Dube, such as:

  * Individuals with histologically confirmed fibrofolliculomas,
  * Individuals with clinical evidence of multiple skin papules consistent with fibrofolliculomas, and/or a family history of spontaneous pneumothorax or kidney cancer
* Individuals with a known germline FLCN mutation
* A relative (related by blood) of an individual with a confirmed or suspected diagnosis of BHD

Design:

* These rare families will be recruited to genetically confirm diagnosis, determine size and location of renal tumors, size at presentation, growth rate and metastatic potential of renal tumors.
* Genetic testing will be offered to gain appreciation of the effect of mutations the BHD gene and to assess the relative activity of various germline and somatic mutations.
* We will determine if there is a relationship between mutation and disease manifestations and phenotype.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Individuals suspected or known to have phenotype or genotype suggestive of Birt-Hogg-Dube, such as:

   * Individuals with at least one histologically confirmed fibrofolliculomas; or
   * Individuals with clinical evidence of multiple skin papules (without fibrofolliculoma biopsy confirmation) and a personal or family history of spontaneous pneumothorax/or kidney cancer; or
   * Individuals with spontaneous pneumothorax and skin papules or kidney cancer and a positive family history of spontaneous pneumothorax, skin papules or kidney cancer; or
   * Individuals with a known germline FLCN gene mutation
2. Renal tumor histology consistent with BHD, including, but not limited to those suggestive of chromophobe, oncocytic neoplasm or oncocytoma.
3. All participants and guardians, for children younger than 18 years of age, must sign an informed consent document indicating their understanding of the investigational nature and the risks of this study before any protocol related studies are performed.
4. Participants must be greater than or equal to 2 years of age.
5. A relative (related by blood) of an individual with a confirmed or suspected diagnosis of BHD.

EXCLUSION CRITERIA:

NONE

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically confirmed fibrofolliculomas, Patients with clinical evidence of multiple skin papules consistent with fibrofolliculomas, and a family history of spontaneous pneumothorax or kidney cancer, a biological relative of a patient with a confirmed diagnosis of BHD. Patients with a known germline FLCN mutation
Sampling Method: Non-Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2002-05-13 (Actual)

PRIMARY OUTCOMES:
Identify genotype / phenotype correlations. | on-going
  Collection of blood, saliva, tissue & urine for Identification of the Disease Gene, and Characterization of the disposition to Renal Cancer
Determine risk of renal cancer, lung cysts and fibrofollicullomas in patients with BHD. | on-going
  Collection of blood, saliva, tissue & urine for Identification of the Disease Gene, and Characterization of the disposition to Renal Cancer
Determine if other genes contribute to BHD. | on-going
  Collection of blood, saliva, tissue & urine for Identification of the Disease Gene, and Characterization of the disposition to Renal Cancer
Define types and characteristics (including patterns of growth) of renal cancer associated with BHD. | on-going
  Collection of blood, saliva, tissue & urine for Identification of the Disease Gene, and Characterization of the disposition to Renal Cancer
Define the natural history of BHD related renal tumors. | on-going
  Collection of blood, saliva, tissue & urine for Identification of the Disease Gene, and Characterization of the disposition to Renal Cancer

CONTACTS AND LOCATIONS:
Overall Officials: W. Marston Linehan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2002-C-0159.html